CLINICAL TRIAL: NCT01126606
Title: Single Center, Open, Cross-over, Phase III Study for Safety and Efficacy (Subjective and Instrumental) Comparative Evaluation Between Dermacyd Silver and Glycerine Vegetal Soap Granado Traditional for Intimate Use in Menopauses Woman.
Brief Title: Comparative Safety and Efficacy Evaluation Between Dermacyd Silver and Glycerine Vegetal Soap Granado Traditional
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LACAC_L_04937
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-12

CONDITIONS: Hygiene
MeSH Terms: interventions — Lactic Acid

ARMS (2):
- Group 1 (Experimental): Dermacyd Silver Frutal followed by Dermacyd Silver Frutal+PH_DESYLSTY_FR followed by wash out followed by Glycerine Vegetal Soap Granado Traditional
  Interventions: Drug: Dermacid Silver (Lactic acid); Drug: Glycerine Vegetal Soap Granado Traditional
- Group 2 (Experimental): Glycerine Vegetal Soap Granado Traditional followed by wash out followed by Dermacyd Silver Floral followed by Dermacyd Silver Floral + PH_DESYLSTY_FR
  Interventions: Drug: Dermacid Silver (Lactic acid); Drug: Glycerine Vegetal Soap Granado Traditional

INTERVENTIONS:
Drug: Dermacid Silver (Lactic acid) — Liquid soap, daily use
Drug: Glycerine Vegetal Soap Granado Traditional — Vegetal soap, daily use

SUMMARY:
Primary Objective:

To evaluate the potential of hydratation and renewal of the mucosa, through corneometry measurement and individual questionnaire perception.

Secondary Objective:

To evaluate the safety in normal condition of use.

ELIGIBILITY:
Inclusion criteria:

* Active sex life
* Menopause for at least 6 months
* Perfect mucosa in the evaluated area
* Use the same cosmetics category

Exclusion criteria:

* Use of antiinflammatory / immunosuppression / antihistaminic drugs
* Personal history of atopy to cosmetic products
* Cutaneous active disease (local and/or general) in the evaluated area
* Disease which can cause immunosuppression, such as diabetes, HIV
* Endocrine pathology such as thyroid disease, ovarian disorder or adrenal gland
* Intense solar exposure (to get a tan) during the 15 days before the evaluation
* Gynaecologic treatment until four weeks before the evaluation
* Whatever vaginal infection detected at time of inclusion
* Other conditions considered by the investigator as reasonable to exclude the patient from the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Transepidermal water loss measurement (TEWL) and corneometry | Up to Week 9
  Measures taken at all visits by Tewameter equipment TM 300. The value of the average will be considered for analysis of final results.
  Corneometry: Measures taken at all visits by Corneometer equipment MPA 580.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil